CLINICAL TRIAL: NCT03499691
Title: An Open-label, Prospective, Randomized, Parallel-Group, Exploratory Study to Explore the Safety and Efficacy of the HDx Therapy Using Theranova 500 Dialyzer in Comparison to Hemodiafiltration
Brief Title: Exploratory Study to Explore the Safety and Efficacy of the HDx Therapy Using Theranova 500 Dialyzer in Comparison to Hemodiafiltration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BXU012191
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Hemodiafiltration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expanded Hemodialysis (HDx) Therapy (Experimental): Patients will undergo 3 dialysis sessions per week with Theranova 500 for up to 24 weeks.
  Interventions: Device: Theranova 500 medium cut-off dialyzer
- Hemodiafiltration (HDF) Therapy (Active Comparator): Patients will undergo 3 dialysis sessions per week with on-line HDF for up to 24 weeks.
  Interventions: Device: Hemodiafiltration

INTERVENTIONS:
Device: Theranova 500 medium cut-off dialyzer — The patients randomized in this group using the Theranova 500 medium cut-off dialyzer, and blood flow rate and treatment duration will be maintained stable during the observation period. However, other prescriptions will vary based on the Principal Investigator's (PI's) judgment. If other dialyzers need to be temporarily used during the study period it shall be recorded which alternative dialyzers are used and for how long the study patient is on a different dialyzer. However, prior to Week 12 laboratory assessment it is recommended that the patient undergoes three dialysis sessions on the designated treatment mode.
  Arms: Expanded Hemodialysis (HDx) Therapy
Device: Hemodiafiltration — The patients randomized in this group using the on-line high-flux HDF dialyzer, in post dilution mode, will continue to receive treatments according to their current treatment prescriptions for the duration of the study.
  Arms: Hemodiafiltration (HDF) Therapy

SUMMARY:
Today it is well established that middle molecules comprise several compounds that are not effectively removed by high-flux dialyzers, and effective clearance of large middle molecules in the process of dialysis depends on the dialyzer membrane having large enough pore sizes, larger than the conventional high-flux dialyzers. Studies have found associations between levels of large middle molecule uremic toxins and immune dysfunction and inflammation, as well as adverse outcomes. This indicates that dialysis membranes having larger pores, enabling an expanded HD (HDx) with more effective removal of large middle molecules, can have a positive impact on the inflammatory state. While data is starting to appear on the long-term use of the HDx therapy, little is still known on how large middle molecules and inflammation markers are affected over time.

ELIGIBILITY:
Inclusion Criteria:

* ESRD patients age between 18 - 80 years
* Clinically stable as judged by the treating physician for 30 days prior to enrollment, as demonstrated by pertinent patient medical history, physical examination, and laboratory testing
* Hemodialysis therapy with HDF for at least 3 months immediately prior to study enrollment

Exclusion Criteria:

* No informed consent provided
* Significant psychiatric disorder, mental disability, or other condition that may interfere with the patient's ability to provide informed consent
* Pregnant, breastfeeding, or planning to become pregnant
* Unstable vascular access associated with risk of low and variable extracorporeal blood flow rate (QB)
* Chronic liver disease, known paraprotein-associated disease, known bleeding disorders (e.g., gastrointestinal bleed, colonic polyps, small bowel angiodysplasia and active peptic ulcers)
* Major bleeding episode (i.e. soft tissue bleeding, blood in stool, joint damage, retinal bleeding, extensive mucosal bleeding, exsanguination, cerebral hemorrhage) ≤ 12 weeks prior to enrollment
* Blood (red blood cell) transfusion ≤ 12 weeks prior to enrollment
* Clinical signs of acute infection ≤ 4 weeks prior to enrollment
* Active cancer, except for basal cell or squamous cell skin cancer
* Positive serology test for human immunodeficiency virus or hepatitis infection
* Scheduled for planned interventions requiring hospitalization > 1 week
* Scheduled for living-donor transplantation within the study period
* Currently participating in another interventional clinical study or has participated in another interventional clinical study in the past 3 months that may interfere with this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2018-10-04 (Actual)

PRIMARY OUTCOMES:
Reduction ratios of lambda immunoglobulin free light chains (λ-FLC) | Week 12
Reduction ratios of kappa immunoglobulin free light chains (k-FLC) | Week 12
Reduction ratios of chitinase-3-like protein 1 (YKL-40) | Week 12
Reduction ratios of fibroblast growth factor 23 (FGF-23) | Week 12
Reduction ratios of serum beta-2 microglobulin (β2M) | Week 12

SECONDARY OUTCOMES:
Change from baseline in mid-week pre-dialysis serum levels of λ-FLC, κ-FLC, YKL-40, FGF-23, ß2M | Week 12 and 24
Change from baseline in mid-week pre-dialysis serum levels of pentraxin-3 (PTX-3), high sensitivity C-reactive protein (hs-CRP), interleukin (IL-6), and interleukin-10 (IL-10) | Week 12 and 24
Percent change from pre- to post-dialysis in mid-week serum levels of hs-CRP | Week 12
Percent change from pre- to post-dialysis in mid-week serum levels of PTX-3 | Week 12
Percent change from pre- to post-dialysis in mid-week serum levels of IL-6 | Week 12
Percent change from pre- to post-dialysis in mid-week serum levels of IL-10 | Week 12
Change from baseline in mid-week pre-dialysis serum level of fibrinogen | Week 12 and 24
Change from baseline in mid-week pre-dialysis serum level of albumin | Week 12 and 24
Single pool Kt/Vurea | Week 24
Serum phosphorous | Week 24
Kidney Disease Quality of Life 36 (KDQOL-36) | Baseline, Week 12, Week 24
Dialysis Symptom Index (DSI) | Baseline, Week 12, Week 24
Serum ferritin | Baseline, Week 12, Week 24
Transferrin Saturation (TSAT) | Baseline, Week 12, Week 24
24-hour urine output on monthly basis | Month 1, Month 2, Month 3, Month 4, Month 5, Month 6
Erythropoiesis stimulating agent (ESA) responsiveness | Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24
Hemoglobin levels | Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24
ESA dosage by type, administration frequency, and route | Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24
Intravenous iron dosage | Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24
Number of adverse events of hospitalization, cardiovascular events, and infective episodes | Week 1 through Week 24
Total patient death | Week 1 through Week 24

CONTACTS AND LOCATIONS:
Locations (1):
- RTS Murcia VII, RTS Servicios de Diálisis S.L.U., Murcia, Spain

REFERENCES:
- [Result] Hadad-Arrascue F, Nilsson LG, Rivera AS, Bernardo AA, Cabezuelo Romero JB. Expanded hemodialysis as effective alternative to on-line hemodiafiltration: A randomized mid-term clinical trial. Ther Apher Dial. 2022 Feb;26(1):37-44. doi: 10.1111/1744-9987.13700. Epub 2021 Jun 29. PMID 34125503